CLINICAL TRIAL: NCT00618592
Title: Does Pre-operative Carbohydrate Loading Reduce Insulin Resistance and Improve Outcomes in Elective Surgical Patients?
Acronym: Preop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: C. David Mazer, St. Michael's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB 02-117
Record Dates: First submitted 2008-02-08; First posted 2008-02-20 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2009-02

CONDITIONS: Coronary Artery Bypass Graft Surgery; Spine Surgery
Keywords: carbohydrate supplementation; cardiac surgery; spine surgery; insulin resistance; insulin sensitivity; short insulin tolerance test; HOMA; outcomes
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CHO (Experimental)
  Interventions: Dietary Supplement: PreOp carbohydrate drink
- FAST (No Intervention)

INTERVENTIONS:
Dietary Supplement: PreOp carbohydrate drink — 800 mL of PreOp evening before surgery, 400 mL at least two hours before surgery
  Other Names: PreOp, Nutricia
  Arms: CHO

SUMMARY:
The recent development of an oral carbohydrate drink for consumption prior to elective surgical procedures has been shown to improve insulin sensitivity. However, these studies have not investigated the use of this carbohydrate supplement in patients undergoing cardiac and spinal surgery.

Hypothesis: The administration of 100g of carbohydrates the evening before and 50g of carbohydrates two hours before elective coronary artery bypass graft (CABG) or spinal surgery will reduce postoperative insulin resistance by 40% compared to those undergoing the standard of care of fasting the evening before and the day of surgery.

DETAILED DESCRIPTION:
In many Western hospitals, including St. Michael's Hospital, fasting for 12-14 hours is the standard protocol for patients entering elective surgery. Fasting results in a depletion of energy stores and consequently, a patient enters surgery in a catabolic state. Furthermore, the human body reacts to surgery by producing a variety of stress hormones and other hormone-like proteins that enable the body to react to stress or injury appropriately. One of the changes that occurs with surgery is related to how the body stores and metabolizes glucose. During and after surgery, muscle and adipose tissue become less sensitive to the action of insulin (insulin resistant). Insulin resistance results in a reduced uptake of glucose by these tissues and subsequently to a rise in circulating blood glucose levels. Sustained high levels of blood glucose have been associated with post-surgical complications and less favourable outcomes. Previous studies have found that fasting before surgery exacerbates insulin resistance during and after surgery. The recent development of a carbohydrate drink for consumption prior to elective surgical procedures has been shown to be well tolerated and pose no additional risk of pulmonary aspiration when ingested two hours prior to surgery. Furthermore, there appears to be metabolic, psychological and possibly clinical benefits in pre-operative carbohydrate loading compared to fasting, including improvements in insulin resistance. However, the studies done to date have been limited by their small sample size, their lack of clinical outcome data and their reliance upon predominantly surgeries of shorter duration and reduced metabolic stress where insulin resistance is lower. Therefore, there is a need to investigate the effect of carbohydrate loading on insulin resistance and clinical outcomes in patients undergoing surgery of extended duration and complexity.

Patients undergoing major cardiac and spinal surgery are ideal for studying the effects of pre-operative carbohydrate loading since this type of operation is of long duration and relatively high surgical stress resulting in the development of significant insulin resistance, and thus potentially benefit from pre-operative carbohydrate loading. Therefore, we will be conducting a larger randomized trial investigating the effects of pre-operative carbohydrate loading in comparison with fasting on insulin resistance and clinical outcomes in patients undergoing invasive cardiac and spinal surgery at St. Michael's Hospital.

We hypothesize that consumption of a pre-operative carbohydrate load will reduce postoperative insulin resistance by 40% (measured by the standardized short insulin tolerance test). As secondary outcomes, we hypothesize that pre-operative carbohydrate loading will reduce circulating markers of inflammation and stress as well as improve clinical outcomes such as blood product utilization, incidence of hyperglycemia, rates of adverse events and length of stay in comparison with standard pre-operative fasting. This study will provide important information regarding the clinical benefits associated with the consumption of a pre-operative carbohydrate load. Many European centres have already liberalized their pre-operative treatments; this study will help to optimize the perioperative management and outcomes of surgical patients at our institution.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing elective coronary artery bypass graft or spinal (decompression and fusion) surgery
* Ability to provide informed consent

Exclusion Criteria:

* Patients undergoing associated cardiac procedures such as valve replacement or valve repair
* Patients undergoing spinal surgery without fusion
* Conditions likely to impair gastrointestinal motility or enhance gastrointestinal reflux
* On medications likely to delay gastric emptying
* BMI > 40
* Existing Type I or Type II diabetes
* Participated in another study in the past 30 days
* Entering surgery greater than five hours after ingestion of morning drink

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | baseline and postoperatively

SECONDARY OUTCOMES:
Markers of inflammation e.g., CRP, IL-6, free fatty acids | baseline, in ICU, and 24, 48 and 72 hours postoperatively
Glucose metabolism e.g., insulin-mediated glucose uptake and GLUT 4 translocation | onset of surgery
Clinical outcomes e.g., length of stay in ICU and hospital, blood transfusions | during surgery and postoperatively
Preoperative patient discomfort | baseline and preoperatively
IGF-1 | baseline, in ICU and 24, 48 and 72 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: C. David Mazer, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Tran S, Wolever TM, Errett LE, Ahn H, Mazer CD, Keith M. Preoperative carbohydrate loading in patients undergoing coronary artery bypass or spinal surgery. Anesth Analg. 2013 Aug;117(2):305-13. doi: 10.1213/ANE.0b013e318295e8d1. Epub 2013 Jun 11. PMID 23757474